CLINICAL TRIAL: NCT04476576
Title: Aerobic Physical Exercise is Cardio-protective in Subjects With Hemato-oncological Disease and New-onset Chemotherapy
Brief Title: Aerobic Exercise is Cardio-protective in Hemato-oncological Disease and New-onset Chemotherapy
Acronym: AEROHEMONCO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucía Florio (Other)
Responsible Party: Sponsor-Investigator, Lucía Florio, Associate Professor Cardiology, Universidad de la Republica
Organization: Universidad de la Republica (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: exercise and chemotherapy
Record Dates: First submitted 2020-07-07; First posted 2020-07-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Cardiotoxicity; Systolic Dysfunction; Exercise, Aerobic
Keywords: cardiotoxicity; systolic dysfunction; exercise, aerobic; chemotherapy; strain
MeSH Terms: conditions — Cardiotoxicity; Motor Activity; Sprains and Strains | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Active group: 3 months , 3 times/week aerobic program Control group: 3 months, 3 times/week flexibility program
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both programs are equally planned related with time and number of sessions as well as clinical monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic (Experimental): 3 months program, 3 times/week aerobic ambulatory program.
  Interventions: Behavioral: Aerobic exercise (experimental)
- Flexibility (Active Comparator): 3 months program, 3 times/week flexibility ambulatory program
  Interventions: Behavioral: Flexibility exercise (active comparator)

INTERVENTIONS:
Behavioral: Aerobic exercise (experimental) — 3 times per week, 30 minutes each time. Entrance in heat: 8-10 min of joint mobility and / or the aerobic exercise in the main part at light intensity (OMNI 3-4) Main part: minimum 30 minutes, maximun 60 minutes. Intensity: moderate, guided by Talk Test and effort perception scale 5-6 OMNI. Type: aerobic, cycling or walking at home using a treadmill or exercise bike and / or cycling and walking outdoors according to the patient's possibilities and preferences. Return to calm: 5 min of aerobic physical activity of main part at mild intensity (OMNI 3-4), then static stretching. Pictures with each type of exercise will be offered and detailed explained.
  Arms: Aerobic
Behavioral: Flexibility exercise (active comparator) — Entrance in heat: 10 min of joint mobility. Main part: Minimum 30 minutes. Frequency: 3 times por week Intensity: The patient should be able to slowly stretch the muscle to a position of mild discomfort. Type: Static Stretch Time: 15-30 seconds 2 repetitions of each stretch Number of exercises: 12 . Pictures with each muscle group to exercise will be offered and detailed explained.
  Arms: Flexibility

SUMMARY:
Oncological diseases are the main cause of death in developed countries and also in Uruguay. Advances in therapeutics have made possible to aspire to cure and in other cases long-term remission with a significant increase in survival and the transformation of cancer into a chronic disease. Chemotherapy treatments have some side effects and cardiotoxicity is well known within them. Heart failure (HF) is a progressive pathology, with high mortality and high resource requirements of the health system with a prognosis that may be worse than some types of cancers. The treatment of established systolic dysfunction and symptomatic HF is mainly based on the indication of inhibitors of the angiotensin-converting enzyme and beta-blockers among other pharmaceutical and no pharmaceutical interventions. Aerobic physical exercise, as a therapeutic intervention, reverses the physiopathological changes that are presumed to lead to HF in sedentary people and it is known, it is feasible to execute an exercise program in cancer patients. However, effective treatments for the primary prevention of systolic dysfunction are not well known. Our hypothesis is that an aerobic physical exercise program for at least 3 months, in subjects with lymphoma and new-onset chemotherapy, is effective in preventing left ventricular systolic dysfunction, at the end of chemotherapy and at one year. For this, the investigators propose a randomized, controlled, clinical study which is blind both for the patient and the evaluating physician, comparing the difference of global longitudinal strain (an echocardiographic result of myocardial function) pre-chemotherapy minus end of chemotherapy and minus one year after, between the active group (aerobic program) and the control group (flexibility program).

DETAILED DESCRIPTION:
Hypothesis: an aerobic physical exercise program for at least 3 months, in subjects with hemato-oncological diseases that initiate chemotherapy, is effective in preventing systolic dysfunction of the left ventricle at the end of chemotherapy and one year.

It is a double-blind, randomized controlled trial. Blinded for the subject, evaluating echocardiographic, and treating hematologist.

Blocked randomization method stratified by sex: the randomization sequence will be software generated and centralized by an investigator independent from assistant physicians and echocardiographic evaluator.

To calculate N sample the investigators took a 15% variation of longitudinal left ventricular strain ( clinically significant criteria). The mean and standard deviation of the healthy Uruguayan population was taken from an own study (19.6 ± 1.7%); considering alpha error 0.05 and power 80%, a sample of 16 in each group is required to find significant results. An additional 20% was added for possible "drop outs" resulting in a sample size of 19 subjects/group (N total 38).

The intervention is a 3 months aerobic exercise program compared with a 3 months flexibility exercise program.

The main outcome is the myocardial longitudinal strain variation. Secondary outcomes are related to systolic and diastolic cardiac function, quality of life, cardiac and oncological outcomes, and evaluation of adherence.

Statistical analysis: Qualitative variables will be expressed in absolute and relative frequency. Continuous variables will be resumed as mean and standard deviation or median and interquartile interval regarding normal distribution. Parametric or non- parametric tests of the association will be used regarding test of normality of each continuous outcome and Chi-squared test for the association of qualitative variables. Survival analysis will be made with Kaplan Meier curves and long rank test.

The project is registered in Uruguayan interventional trial registration (Ministery of Public Health) with the number 812559.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years old
* New-onset chemotherapy
* Lymphoma (Hodgkin or non-Hodgkin).

Exclusion Criteria:

* Inability or contraindication to moderate physical activity due to orthopedic cause or general disease (excluding oncological).
* Hemato-oncological pathology different from lymphomas.
* Lymphomas not treated with anthracyclines
* Non-sinus rhythm.
* Poor echocardiographic window (inability to assess longitudinal strain in more than 4 segments).
* Physically active subjects (practice aerobic exercise at least 30 minutes, 3 times / week, 3 previous months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in GLS (exercise of flexibility and balance). | 6 months
  GLS will be measured as the mean value of all segments pick systolic longitudinal strain expressed in percentage (%). The method will be speckle tracking, with a 4 MHz traducer and ViviIQ General Electric echocardiographer, The difference between GLS pre Chemotherapy minus post-chemotherapy and GLS pre chemotherapy minus a year after.

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 1 year
  LVEF evaluated through Simpson biplane method, expressed in percentage. The value to compare will be those at the end of chemotherapy and a year after the beginning.
GLS | 1 year
  GLS evaluated through speckle tracking method, expressed in percentage. The value to compare will be those at the end of chemotherapy and a year after the beginning.
Cardiotoxicity incidense | 1 year
  Cardiotoxicity definition: Decline of 10% or more of LVEF (pre chemotherapy value is the reference). Incidence of cardiotoxicity will be compared at the end of chemotherapy and one year after.
Diastolic function. E/e´index | 1 year
  Pick value of E wave (pulse Doppler at the tip of mitral valve, first positive wave) and pick value of e´(mean of basal septal and basal lateral e´ , evaluated with tissue Doppler). The comparison will be done at the end of chemotherapy and 1 year from the beginning.
Diastolic function. Left atrial GLS | 1 year
  Biplane atrial GLS expressed in percentage (%). Method for estimation: speckle tracking. The comparison will be at the end of chemotherapy and 1 year from the beginning.
Diastolic function. Left atrial volume. | 1 year
  Biplane left atrial volume, through longitud-area method, expressed in ml. The comparison will be at the end of chemotherapy and 1 year from the beginning.
Cardiac injury. Troponin I dosification. | 3 months
  Dosification of troponin I value (ng/ml) between groups (data from Day 8 to 11 of third chem cycle)
Clinical cardiovascular composite outcome | 1 year
  Incidence of HF incomes and cardiovascular mortality during the follow-up year between groups. Comparison of survival free of events (Kaplan Meier curve and long rank test).
Muscle corporal mass | 1 year
  Percentage of muscle mass calculated through a bioimpedance balance. Comparison will be made baseline, at 3 months and a year.
Physical activity. Monthly mean of steps. | 3 months
  The monthly average of daily physical activity during the 3 months duration of the exercise program measured by steps of a physical activity wristband.
Quality of life. Minnesota LIVING WITH HEART FAILURE® Questionnaire (MLHFQ) | 3 months
  Minnesota questionnaire for HF patients: It is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. The patient marks a 0 (zero) to 5 scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses. The response format ranges from 0 (none or not applicable), to 1(very little) to 5 (very much). The simple sum of the responses that ranges from 0 to 105 is a measurement of heart failure severity as indicated by its adverse effect on the respondent's life during the past month. The MLHFQ scores increase with the adverse impact of heart failure on the respondent's life. Evaluation made at the end of exercise program.
Quality of life. Functional Assessment of Cancer Therapy (FACT) | 3 months
  FACT-G (general) questionnaire for oncological patients.General quality of life instrument intended for use with a variety of chronic illness conditions. Originally validated in a general cancer population.Administration: Self Time to complete: 5 minutes. Number of items:27 Domains & categories: 4 Name of categories/domains: Physical, social/family, emotional, and functional well-being. Scaling of items: Five-point scale from 0 (not at all) to 4 (very much). Evaluation made at the end of exercise program.
Dysnea | 3 months
  PROMIS questionnarie for dysnea severity evaluation.The PROMIS Dyspnea Severity item bank assesses the severity of shortness of breath or difficulty breathing an adult experiences in response to various specific activities. Each activity is rated in terms of degree of dyspnea (no shortness of breath, mildly short of breath, moderately short of breath, severely short of breath) while engaging in the activity over the past 7 days, with higher scores reflecting greater levels of dyspnea. Respondents who indicate that they did not perform an activity in the past 7 days will not produce a score for that item. The bank includes 33 items.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Florio, MD MSc, Principal Investigator — Universidad de la Republica
Locations (1):
- Centro Cardiovascular Universitario-Hospital de Clínicas -FMED- UdelaR, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No